CLINICAL TRIAL: NCT04085354
Title: Evaluation of the Clinical Efficacy and Safety of Dapoxetine, Combined Dapoxetine With Folic Acid and Combined Dapoxetine With Vitamin B12 in Treatment of Patients With Premature Ejaculation: A Randomized Placebo-controlled Clinical Trial
Brief Title: Evaluation of the Clinical Efficacy and Safety of Dapoxetine, Combined Dapoxetine With Folic Acid and Combined Dapoxetine With Vitamin B12 in Treatment of Patients With Premature Ejaculation
Acronym: PE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abu El-Hamd, Assistant Professor of Dermatology, Venereology and Andrology Department, Faculty of Medicine, Sohag University, Egypt., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2019
Record Dates: First submitted 2019-08-30; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Geritol; dapoxetine; Folic Acid; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: All patients will be randomized equally divided into four groups (30 patients each).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The distribution of the patients among the four groups was based on randomized coded cards, so the patients were unaware of the type of the drugs used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Group 1 was given placebo in form oral multivitamin tablet 1 h before intercourse.
  Interventions: Drug: Multi-Vitamin Tablets
- Dapoxetine (Active Comparator): Group 2 was given on-demand 30 mg dapoxetine 1-2 h before intercourse.
  Interventions: Drug: Dapoxetine
- Dapoxetine and folic acid. (Active Comparator): Group 3 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg folic acid.
  Interventions: Drug: Dapoxetine and folic acid.
- Dapoxetine and vitamin B12 (Active Comparator): Group 4 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg vitamin B12
  Interventions: Drug: Dapoxetine and vitamin B12

INTERVENTIONS:
Drug: Multi-Vitamin Tablets — The distribution of the patients among the four groups was based on randomized coded cards, so the patients were unaware of the type of the drugs used. Group 1 was given placebo in form oral multivitamin tablet 1 h before intercourse.
  Arms: Placebo
Drug: Dapoxetine — The distribution of the patients among the four groups was based on randomized coded cards, so the patients were unaware of the type of the drugs used. Group 2 was given on-demand 30 mg dapoxetine 1-2 h before intercourse.
  Arms: Dapoxetine
Drug: Dapoxetine and folic acid. — The distribution of the patients among the four groups was based on randomized coded cards, so the patients were unaware of the type of the drugs used. Group 3 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg folic acid.
  Arms: Dapoxetine and folic acid.
Drug: Dapoxetine and vitamin B12 — The distribution of the patients among the four groups was based on randomized coded cards, so the patients were unaware of the type of the drugs used. Group 1 was given placebo in form oral multivitamin tablet 1 h before intercourse. Group 4 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg vitamin B12
  Arms: Dapoxetine and vitamin B12

SUMMARY:
This study will aim to assess of the clinical efficacy and safety of dapoxetine, combined dapoxetine with folic acid and combined dapoxetine with vitamin B12 in treatment of patients with premature ejaculation: A randomized placebo-controlled clinical trial.

DETAILED DESCRIPTION:
In a single-blind placebo-controlled clinical study, it will be carried out on 120 patients with PE.

All patients will be randomized equally divided into four groups (30 patients each).

Group 1 was given placebo in form oral multivitamin tablet 1 h before intercourse.

Group 2 was given on-demand 30 mg dapoxetine 1-2 h before intercourse. Group 3 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg folic acid.

Group 4 was given on-demand 30 mg dapoxetine 1-2 h before intercourse and daily oral supplementation of 0.5 mg vitamin B12

ELIGIBILITY:
Inclusion Criteria:

Premature ejaculation

Exclusion Criteria:

* Erectile dysfunction
* Diabetes mellitus
* chronic prostatitis
* Advanced renal or hepatic diseases
* Neurological diseases

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Arabic Index of Premature Ejaculation | 0-6 weeks after treatment
  The AIPE questionnaire includes seven questions.Response to each question will be scored on a scale from 1 to 5.
Intravaginal ejaculatory latency times | 0-6 weeks after treatment
  By using stopwatches

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abu El-Hamd, MD, Principal Investigator — Assistant Professor
Locations (1):
- Faculty of Medicine, Sohag University, Egypt, Sohag, Egypt